CLINICAL TRIAL: NCT06289816
Title: Minimally Invasive Spleen Preserving Surgery to Treat Primary Splenic Hydatidosis: Short and Long Term Outcomes: A Cohort Study
Brief Title: Spleen Preserving Surgery for Splenic Hydatidosis: A Cohort Study on Short and Long-Term Outcomes
Status: Completed | Type: Observational
Sponsor: Yarmouk University (Other)
Responsible Party: Principal Investigator, Anas Aljaiuossi, Consultant Hepatobiliary Surgeon, Yarmouk University
Other Study IDs: 28/01/2023
Record Dates: First submitted 2024-02-24; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Spleen-Preserving Surgery; Echinococcus Granulosus Infection; Hydatid Disease; Minimally Invasive Surgery
Keywords: Spleen-Preserving Surgery; Primary Splenic Hydatid Cyst; Hydatid Disease; Minimally Invasive Surgery; Echinococcus granulosus; Recurrence
MeSH Terms: conditions — Echinococcosis; Recurrence | interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Minimally Invasive Surgery — Minimally Invasive Surgery : Laparoscopic partial splenectomy, cystectomy, and cyst deroofing.

SUMMARY:
This retrospective cohort study examines the effectiveness of minimally invasive spleen-preserving surgeries compared to total splenectomy for treating primary splenic hydatidosis in Jordan. Covering 18 patients from January 2015 to June 2021, the research highlights similar recurrence rates between both surgical approaches, emphasizing the benefits of spleen preservation in maintaining immune function and reducing septic risks, particularly in pediatric patients.

DETAILED DESCRIPTION:
The study delves into a detailed analysis of 18 cases of primary splenic hydatid cysts treated through spleen-preserving surgeries-laparoscopic partial splenectomy, cystectomy, and cyst deroofing-augmented by albendazole therapy. It presents a comprehensive comparison based on patient demographics, symptoms, surgical details, and outcomes, including complications and recurrence rates. Findings reveal no significant statistical difference in recurrence rates between spleen-preserving methods and total splenectomy, suggesting the viability of less invasive approaches for managing this condition effectively while preserving spleen functionality and minimizing post-operative complications. The study underlines the need for individualized treatment plans and further research with larger cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 14 years or older).
* Diagnosed exclusively with primary, non-recurrent splenic hydatid cysts.

Exclusion Criteria:

* Children under 14 years of age.
* Patients in late pregnancy.
* Individuals with recurrent cysts.
* Cases with extra-splenic involvement.
* Patients with less than two years of postoperative follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study involved patients diagnosed with primary splenic hydatid cysts, from January 2015 to June 2021. The study included medical records of 18 patients aged 14 years or older, diagnosed exclusively with primary, non-recurrent splenic hydatid cysts.
  Exclusion criteria encompassed individuals under 14 years, patients in late pregnancy, those with recurrent cysts, extra-splenic involvement, or less than two years of postoperative follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Postoperative Short-Term Complications | Up to 1 month post-operation
  The measure focuses on the incidence and nature of short-term complications following spleen-preserving surgeries compared to total splenectomy. Short-term complications may include infection, bleeding, or any other immediate post-surgical issues that impact recovery.
Incidence of Postoperative Long-Term Complications | Up to 2 years post-operation
  This measure assesses the long-term complications associated with spleen-preserving surgeries versus total splenectomy. Specifically, it examines the recurrence of hydatid cysts as a significant long-term complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Anas Aljaiuossi, Irbid, Jordan